CLINICAL TRIAL: NCT05252650
Title: Postoperative Pain Management in Pediatric Patients With Cerebral Palsy - Comparative Observational Study"
Brief Title: Postoperative Pain Management in Cerebral Palsy - Comparative Observational Study"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, investigator, Biruni University
Other Study IDs: biruni cp
Record Dates: First submitted 2022-02-13; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- regional block: epidural / peripheral nerve block
  Interventions: Behavioral: pain
- intravenous: intravenous analgesia
  Interventions: Behavioral: pain

INTERVENTIONS:
Behavioral: pain — postoperative pain

SUMMARY:
In this study, our aim is to examine orthopedic interventions, anesthesia method, postoperative pain level and management applied to patients with CP in biruni university hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral palsy between the ages of 3-15,
* Category 2 according to the Classification of the American Society of Anesthesiology (ASA 2),
* patients undergoing soft tissue release for knee or ankle flexion contracture of the lower extremity with palliative or reconstructive hip interventions

Exclusion Criteria:

* Any child with CP younger than 3 years old and older than 15 years has undergone
* procedures without a specific diagnosis of CP,
* the need for bone surgery,
* requiring both hip, knee and ankle surgery in the same session,
* with autonomic neuropathy,
* Patients with a history of anticholinergic and vasoactive drug use or allergy to amide type local anesthetics

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 130 patients aged 3-15 years with a diagnosis of cerebral palsy, category 2 according to the Classification of the American Society of Anesthesiology (ASA 2), who underwent soft tissue release for knee or ankle flexion contracture of the lower extremity with palliative or reconstructive hip interventions
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2022-07-28 (Estimated); Study Completion 2022-08-05 (Estimated)

PRIMARY OUTCOMES:
pain score | 6 month
  pain score with r-FLACC

CONTACTS AND LOCATIONS:
Locations (1):
- Ilke Kupeli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kim SH, Chun DH, Chang CH, Kim TW, Kim YM, Shin YS. Effect of caudal block on sevoflurane requirement for lower limb surgery in children with cerebral palsy. Paediatr Anaesth. 2011 Apr;21(4):394-8. doi: 10.1111/j.1460-9592.2011.03530.x. Epub 2011 Feb 8. PMID 21299684
- [Result] Ozkan D, Gonen E, Akkaya T, Bakir M. Popliteal block for lower limb surgery in children with cerebral palsy: effect on sevoflurane consumption and postoperative pain (a randomized, double-blinded, controlled trial). J Anesth. 2017 Jun;31(3):358-364. doi: 10.1007/s00540-017-2318-2. Epub 2017 Feb 14. PMID 28197774
- [Result] Evreinov, V. V., & Zhirova, T. A. (2020). Regional anesthetic techniques for hip surgery in children with cerebral palsy. Genij Ortopedii, 26(4), 521-256.
- [Result] Pedersen LK, Rahbek O, Nikolajsen L, Moller-Madsen B. The revised FLACC score: Reliability and validation for pain assessment in children with cerebral palsy. Scand J Pain. 2015 Oct 1;9(1):57-61. doi: 10.1016/j.sjpain.2015.06.007. PMID 29911640